CLINICAL TRIAL: NCT06408948
Title: Phase I Clinical Trial of Mass Balance of [14C]SHR7280 in Healthy Chinese Subjects
Brief Title: A Study to Evaluate the Mass Balance of [14C]SHR7280 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SHR7280-106
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Assisted Reproduction

STUDY DESIGN:
Intervention Model Description: Single oral dose of [14C]SHR7280
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]SHR7280 (Experimental)
  Interventions: Drug: [14C]SHR7280

INTERVENTIONS:
Drug: [14C]SHR7280 — Patients will receive single dose of orally [14C]SHR7280 on Day 1.

SUMMARY:
Evaluate the Mass Balance of [14C]SHR7280 in Healthy Adult Volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form prior to the trial and have a full understanding of the trial's procedures, content, and potential adverse reactions;
2. Healthy adult females and males between 18 and 45 years;
3. Body weight ≥50 kg(for male), body weight ≥45 kg(for female), and the body mass index (BMI) of 19 to 26 kg/m2;
4. From the signing of the informed consent form until 12 months after the last administration, the subject (including partner) has no family planning and is willing to use the high-efficiency contraceptive measures specified in the plan;
5. The first three menstrual cycles for women were regular, with a menstrual cycle of 21-35 days, and no abnormal uterine bleeding occurred.

Exclusion Criteria:

1. Comprehensive physical examination, vital signs, laboratory tests (blood routine, blood biochemistry, coagulation function, urine analysis, fecal routine+occult blood, thyroid function), full chest X-ray, 12 lead electrocardiogram, abdominal ultrasound, digital rectal examination, bilateral breast, uterus, and bilateral accessory ultrasound results that the researcher deems clinically significant;
2. Serum testosterone (T) <3.46 ng/mL during screening for male; serum follicle stimulating hormone (FSH) ≥ 25mIU/mL during screening period for female;
3. Patients with QTcF>450 msec (male) and QTcF>470 msec (female) at the time of screening or baseline, or other clinically significant abnormalities determined by the researcher;
4. Hepatitis B surface antigen (HBsAg) positive, or anti hepatitis C virus (HCV) antibody positive, or human immunodeficiency virus (HIV) antigen/antibody combined test positive, or Treponema pallidum antibody positive;
5. Screening period or baseline period (D-1) serum pregnancy testing (serum β- The HCG test )result is positive for female;
6. Women use the following contraceptive methods during screening visits: sustained-release intrauterine devices, sustained-release contraceptives (subcutaneous implants, vaginal rings, microspheres, and microcapsules); Before screening, use long-acting contraceptive pills (using medroxyprogesterone acetate for 3 months and other injections for 1 month), oral contraceptives (such as short acting, long-acting, or emergency contraceptives) for 2 months before screening, and contraceptive patches for 1 month before screening; Special circumstances to be determined by the researcher;
7. Abuse of drugs or use of soft drugs (such as marijuana) in the three months prior to screening, or use of hard drugs (such as amphetamines, phencyclidine, etc.) in the year prior to screening; Or screening period urine drug test positive individuals, including: morphine, methamphetamine (methamphetamine), ketamine, ecstasy (methamphetamine), marijuana (tetrahydrocannabidiol acid);
8. Using any prescription, over-the-counter, herbal or dietary supplements before the first two screening weeks;
9. Women with a history of pregnancy, miscarriage, childbirth, or breastfeeding in the 6 months prior to screening;
10. Any clinical history of serious diseases or conditions that the researcher believes may affect the trial results, including but not limited to a history of circulatory, endocrine, nervous, digestive, urinary, or blood, immune, mental, and metabolic diseases;
11. Individuals with a history of malignant tumors or suspected to have sex hormone dependent malignant tumors;
12. Allergic constitution, or suspected allergy to any ingredient in SHR7280 formulation;
13. Individuals who have undergone any surgery in the first 3 months prior to screening, have not yet recovered after surgery, or are expected to have surgery or hospitalization plans during the trial period;
14. Perianal diseases with hemorrhoids or periodic/ongoing rectal bleeding; The subject is unable to swallow, or has a history of gastrointestinal dysfunction such as irritable bowel syndrome, inflammatory bowel disease, or has undergone surgery such as gastrectomy, which the researcher determines may affect drug absorption;
15. Habitual constipation or diarrhea;
16. Have a history of severe vomiting;
17. Individuals with a history of smoking in the first three months prior to screening (average daily smoking>5 cigarettes);
18. In the three months before screening, the average daily intake of alcohol exceeded 25 g (for example, 750 mL of beer, 250 mL of wine, or 50 mL of Baijiu); Or those with an alcohol breath test result of ≥ 20 mg/dl during the screening period;
19. Habitually drinking grapefruit juice or excessive amounts of tea, coffee, and/or caffeinated beverages, or unable to quit during the trial period;
20. Select clinical trial participants who have participated in any other drug or medical device within the first 3 months or within 5 half-lives of the drug (depending on whether the drug is administered or the device is used);
21. Those who receive the vaccine within 2 weeks before the first administration or within 1 month after the last administration during the study period;
22. Individuals who have donated (or lost) blood and have donated (or lost) more than 400 mL of blood, or have received blood transfusions in the first 3 months prior to screening;
23. Engaged in workers who require long-term exposure to radioactive conditions; Or select individuals who have been significantly exposed to radiation (chest/abdominal CT ≥ 2 times, or other types of X-ray examinations ≥ 3 times) or have participated in radiopharmaceutical labeling trials in the one year prior to screening;
24. Difficulty swallowing, difficulty in venous blood collection, or physical condition unable to withstand blood collection; Or subjects who are expected to be unable to complete the entire trial follow-up;
25. According to the researcher's judgment, the subjects may have factors that affect drug absorption, distribution, metabolism, and excretion, or may reduce compliance, or other factors that are not suitable for participation in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2024-06-07 (Actual); Primary Completion 2024-07-06 (Actual); Study Completion 2024-07-06 (Actual)

PRIMARY OUTCOMES:
Cumulative recovery and recovery rate of total radioactive substance in urine and feces | 0-240 hours
Percentage of parent drug and its metabolites in plasma as a percentage of total radioactive exposure (%AUC) | 0-120 hours
Percentage of parent drug and its metabolites in urine and feces as a percentage of administered dose (%Dose) | 0-240 hours
Radioactivity Tmax | 0-120 hours
Radioactivity Cmax | 0-120 hours
Radioactivity AUC | 0-120 hours
Radioactivity t1/2 | 0-120 hours
Radioactivity CL/F | 0-120 hours
Radioactivity Vz/F | 0-120 hours
Total radioactivity ratio for blood/plasma | 0-48 hours

SECONDARY OUTCOMES:
Plasma SHR7280: Tmax | 0-120 hours
Plasma SHR7280: Cmax | 0-120 hours
Plasma SHR7280: AUC | 0-120 hours
Plasma SHR7280: t1/2 | 0-120 hours
Plasma SHR7280: CL/F | 0-120 hours
Plasma SHR7280: Vz/F | 0-120 hours
Plasma SHR7280: λz | 0-120 hours
AEs and SAEs | Screening to 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided